CLINICAL TRIAL: NCT06710769
Title: Ovarian Tissue Freezing For Fertility Preservation In Girls Facing A Fertility Threatening Medical Diagnosis Or Treatment Regimen
Brief Title: Ovarian Tissue Cryopreservation
Acronym: OTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-195
Record Dates: First submitted 2023-11-06; First posted 2024-11-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: This study is an investigation of the characteristics of patients who utilize ovarian tissue cryopreservation, the timing of ovarian tissue use, and pregnancy outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- girls facing possible infertility (Other): Newly diagnosed female or relapsed malignancy who is 1-25 years of age with proposed treatment regimen containing at least ONE (1) of the following:
  whole abdomen or pelvic irradiation total body irradiation
  Proposed treatment regimen to include any of the following:
  cyclophosphamide equivalent dose (CED, see Green et al 2014) ≥7.5 g/m2 any treatment regimen containing procarbazine bone marrow transplant conditioning regimen containing alkylator OR health condition or malignancy that requires removal of one or both ovaries
  Interventions: Procedure: Ovarian tissue removal will be performed laparoscopically

INTERVENTIONS:
Procedure: Ovarian tissue removal will be performed laparoscopically — under general anesthesia concomitantly with another scheduled procedure if possible. Following removal, ovarian tissue will be shipped to University of Pittsburg Medical Center, Magee-Womens Research Institute for processing. Freezing and storing techniques will be in accordance with FDA regulations for reproductive tissues, guidelines of the American Association of Tissues Banks and any other applicable federal, state and local regulations. The tissue will be carefully separated dividing the cortex from the medulla. The cortex will then be cryopreserved for long term storage. The medulla will be shipped overnight back to the PCH Department of Pathology for histological evaluation. If pathology finds evidence of cancer in the ovarian tissue provided, they may request that all of the patient's tissue be returned to pathology for a more detailed examination, which may eliminate the tissue available for the patient's future use.

SUMMARY:
Ovarian Tissue Freezing For Fertility Preservation In Girls Facing A Fertility Threatening Medical Diagnosis Or Treatment Regimen

DETAILED DESCRIPTION:
Cancer is a health concern; however, science advancement in disease detection and treatment modalities continues to improve patient survival rates. Cancer treatment consequences are gaining importance for survivors, families and providers. Infertility is a primary concern among female cancer survivors as it not only has biological implications, but psychosocial implications as well. Cancer treatment can cause acute ovarian failure, premature menopause and results in reproductive challenges in survivorship. Females who are approaching reproductive age at time of cancer diagnosis, who receive abdominopelvic radiation or high dose alkylating agents and those diagnosed with Hodgkin's lymphoma have increased risk for infertility following treatment. Cancer treatment is not the only treatment that threatens reproductive capacity, but rheumatoid arthritis and lupus treatment may also cause infertility.

Female cancer patients express fertility preservation is extremely important for their long-term psychosocial health. The current American Society for Clinical Oncology Clinical Practice Guideline states that all patients should be made aware of possible side effects of treatment on fertility, and that patients be offered fertility preservation interventions. Embryo banking or egg banking (oocyte preservation) prior to chemotherapy is the most successful options for fertility preservation in women. This option necessitates time for ovarian stimulation and retrieval which can take up to 2-3 weeks and is costly. This option may be longer for those who acquire ovarian hyper-stimulation syndrome and younger patients have a higher risk for OHSS. Embryo banking requires mature oocytes and can cause emotional and physical stress. The financial and physical challenges with fertility preservation motivate the desire to find alternatives for young cancer patients.

Improved freezing and thawing techniques for human oocytes have contributed to pregnancy rates comparable to those using fresh egg following in vitro fertilization. Prior to ovarian tissue cryopreservation there was no fertility preservation intervention available to patients who could not delay treatment or were too young to undergo hormonal stimulation. As of 2017, greater than 130 live births following transplantation of frozen/thawed ovarian tissue have been reported. Ovarian tissue cryopreservation has proven to be a safe and efficient method for preserving future fertility for patients undergoing potentially sterilizing treatments. Ovarian tissue cryopreservation is a standard-of-care in parts of Europe and is routine in several children's hospitals throughout the United States. We propose this option be available to qualifying patients at Phoenix Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed or relapsed malignancy with proposed treatment regimen containing at least ONE (1) of the following:

whole abdomen or pelvic irradiation

total body irradiation

Proposed treatment regimen to include any of the following:

cyclophosphamide equivalent dose (CED, see Green et al 2014) ≥7.5 g/m2

any treatment regimen containing procarbazine

bone marrow transplant conditioning regimen containing alkylators

OR health condition or malignancy that requires removal of one or both ovaries. Health status adequate to undergo elective laparoscopic surgery (as per anesthesiologist assessment)

Exclusion Criteria:

* Pregnancy or a patient who is currently breastfeeding

Patients who are eligible for and agree to oocyte preservation

Anyone deemed high risk for complications from the surgery and/or anesthesia.

Anyone unable to provide consent due to psychiatric conditions or cognitive delay (in parent/guardian for patients <18 years, and patient >18 years)

Ages: 1 Year to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female patients who are facing a fertility threatening diagnosis and/or treatment
Enrollment: 40 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who utilize their ovarian tissue and the age at which they use it will be evaluated. The number of patients who elect to have OTC will be analyzed over time to identify trends. | 10 years
  data will be investigated via qualitative analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Childrens, Phoenix, Arizona, United States